CLINICAL TRIAL: NCT01395290
Title: Vitamin D and Staphylococcus Aureus in the Diabetes Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UIT-ENDO-2011-1
Record Dates: First submitted 2011-07-14; First posted 2011-07-15 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Infection
Keywords: staphylococcus aureus; vitamin D
MeSH Terms: conditions — Infections; Staphylococcal Infections | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- cholecalciferol (Experimental): cholecalciferol 20.000 IU per week
  Interventions: Drug: cholecalciferol

INTERVENTIONS:
Drug: cholecalciferol — 20.000 IU per week, oral

SUMMARY:
There are indications that the vitamin D status of an individual is related to susceptibility to staphylococcal infections. In the present study we will examine nasal colonisation rate in subjects participating in an ongoing vitamin D intervention study ( 20.000 IU cholecalciferol per week vs placebo) for the prevention of type 2 diabetes in subjects with impaired glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* participant in an ongoing intervention study with vitamin D

Exclusion Criteria:

* none specifically for this study

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
nasal staphylococcus colonisation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Jorde, Professor, Principal Investigator — University of Tromso
Locations (1):
- University Hospital of North Norway, Tromsø, Tromsø, Norway